CLINICAL TRIAL: NCT05179980
Title: Design of a Comprehensive Model for the Evaluation of Trustable Professional Activities in the General Surgery Setting
Brief Title: Comprehensive Model for Evaluation of Surgical EPAs
Status: Completed | Type: Observational
Sponsor: Hospital General de Chihuahua - Dr. Salvador Zubirán Anchondo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 00189
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Entrustable Professional Activities
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Evaluation of clinical-surgical competencies with a previously validated instrument.
  Other Names: Evaluation

SUMMARY:
Introduction. Competency-based medical education (CBME) frameworks have become increasingly prevalent among surgical education accreditation bodies. Medical schools, postgraduate training programs, and licensing bodies conduct assessments to certify the competence of future practitioners, and judge the adequacy of training programs.

Methods. A prospective cohort study was designed to evaluate clinical-surgical competencies in all residents of a general surgery program. All medical residents of the general surgery program of the Faculty of Medicine and Biomedical Sciences at the Autonomous University of Chihuahua, were video recorded with consent, in the field (Outpatient consultation, Surgical ward, Inpatient room, Classroom), for posterior evaluation by the professors of the program with electronic rubrics made with Google forms.

DETAILED DESCRIPTION:
A prospective cohort study was designed to evaluate clinical-surgical competencies in residents of the general surgery program during the 2020-2021 academic year at a single, secondary care, public medical institution.

For this purpose a previously validated instrument for the comprehensive evaluation of clinical-surgical competencies was used (9), which considered five dimensions, derived from the Single Plan for Medical Specialties in terms of 1-3) Clinical-surgical care (preoperative, transoperative and postoperative management), 4) Search and transfer of knowledge, and 5) Research proficiency. Each instrument was composed of 6 to 7 items, graduated in four levels of achievement; a) responsive, b) resolutive, c) autonomous, and d) strategic.

All surgery residents were video recorded with consent, in the field (Outpatient consultation, Surgical ward, Inpatient room, Classroom) for posterior self-evaluation, co-evaluation and hetero-evaluation with electronic rubrics made with Google forms.

ELIGIBILITY:
Inclusion Criteria:

* Residents in an universitary general surgery program

Exclusion Criteria:

* Staff surgeons
* Residents from another universitary program

Ages: 23 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of the general surgery program at a secondary care, public medical institution.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Entrustable Professional Activities | 2020-2024 academic years
  Important work tasks that trainees need to be able to perform with supervision at a distance by the end of Basic Training

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Cervantes-Sánchez, MD, MSc, Principal Investigator — Chihuahua City General Hospital "Dr. Salvador Zubirán Anchondo"
Locations (1):
- Chihuahua City General Hospital "Dr. Salvador Zubirán Anchondo", Chihuahua City, Mexico

IPD SHARING:
Plan to Share IPD: No